CLINICAL TRIAL: NCT00793208
Title: Active Immunization of Patients With Non Small Cell Lung Cancer (NSCLC) Using Fibroblasts Transfected With DNA From Autologous Tumor (Phase IB Study)
Brief Title: Immunization of Patients With Non Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: study closed due to low enrollment
Sponsor: Theresa Whiteside, PhD (Other)
Collaborators: Immune Cell Therapy Inc. (Industry)
Responsible Party: Sponsor-Investigator, Theresa Whiteside, PhD, Professor of Pathology,Director of the UPCI IMCPL Facility, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-004
Record Dates: First submitted 2008-11-13; First posted 2008-11-19 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
Keywords: Lung cancer; non small cell; vaccine; carcinoma; immunization; autologous Tumor; vaccination
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Carcinoma | interventions — DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine (Experimental): vaccine composed of lethally irradiated semi-allogeneic human fibroblasts transfected with genomic tumor DNA from the patient's own tumor
  Interventions: Biological: semi-allogeneic human fibroblasts (MRC-5) transfected with DNA

INTERVENTIONS:
Biological: semi-allogeneic human fibroblasts (MRC-5) transfected with DNA — Each vaccine consists of 1 x 10e7 DNA-transfected irradiated fibroblasts. A total of 4 weekly immunizations will be delivered to each patient. Each vaccine will be administered i.d. using a 1 mL syringe and a 25 gauge needle.
  Subjects will have immunizations administered at 4 different sites for each vaccination as follows:
  Site #1: Right arm Site #2: Left arm Site #3: Right thigh Site #4: Left thigh Approximately equal numbers of transfected fibroblasts will be administered at each site.

SUMMARY:
The study of the vaccine will proceed in two stages after the method of Simon (102). In the first stage, 15 patients will be accrued and treated. If two or fewer objective immunologic responses occur, the study will be terminated. If 3 or more responses are observed, the study will proceed to the second stage, accruing an additional 22 patients. If the second stage is complete and a total of 9 or more immunologic responses are observed among the 37 patients treated, the treatment response rate for the vaccine will be considered high enough to warrant further study. Conversely, if the evaluation of the vaccine concludes at the first stage, or if 8 or fewer total immunologic responses occur after completing the second stage, the vaccine will not be considered for further study.

DETAILED DESCRIPTION:
This is an uncontrolled, non-randomized trial to evaluate safety, immunogenicity and feasibility of a new vaccine, consisting of semi-allogeneic fibroblasts transfected with autologous tumor-derived DNA. Briefly, the plan is to use a two-stage trial design and to initially enroll 15 patients with non small cell lung cancer (NSCLC) over a period of 2 years. The patients will undergo surgery and a portion of the primary tumor specimen not necessary for the pathologic diagnosis will be obtained to serve as a source of tumor DNA. Each DNA-based vaccine will contain 1 x 10e7 DNA-transfected human allogeneic fibroblasts. The vaccine will be lethally irradiated before it is used for immunization. It will be administered intradermally in the Outpatient Clinic. Patients delayed-type hypersensitivity (DTH) responses will be tested but will not be an eligibility criterion. Immunologic response to the vaccine will be evaluated. If there is no evidence of toxicity, and >3 of the 15 initial patients show immunologic response, the second stage of the study will be opened for accrual of 22 patients. All patients will be monitored by IFN-g secretion in ELISPOT assays prior to and after vaccination for the frequency of T-cells responsive to autologous tumor (if available) and/or to the vaccine. The patients will also be evaluated before and after vaccination for the capability of their T cells to respond to activating signals delivered via the T cell receptor (TcR).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent conforming to the institutional guidelines obtained from the patient.
* A diagnosis of non-small cell lung cancer (NSCLC), subjects will undergo or have had surgical resection.
* Age 18 or above.
* Karnofsky performance status > 70
* Adequate hematologic function:

  * Absolute neutrophil count > 1,000/mm3
  * Absolute lymphocyte count > 1,000/mm3
  * Hemoglobin > 9 g/dL
  * Platelets > 100,000/mm3
* Liver function tests:

  * Bilirubin (total) < 1.7 mg/dL
  * Alkaline phosphatase < 252 u/L
  * SGOT < 108 u/L
* Kidney profile:

  * Serum electrolytes

    * Sodium 136-146 mEq/L
    * Potassium 3.5-5.0 mEq/L
    * Bicarbonate 21-31 mEq/L
    * Chloride 98-107 mmol/L
  * Serum creatinine < 3 x ULN
  * BUN 8-26 mg/dL
* At least a 12 week interval should have elapsed between vaccination and any prior radiation therapy, chemotherapy or any other treatment. Patients should have recovered from surgery and adjuvant treatment.

Exclusion Criteria:

Subjects will be EXCLUDED from participation in the study if any of the following apply:

* One or more of the Inclusion Criteria are not met.
* A significant history or current evidence of cardiac disease including, but not limited to: congestive heart failure, coronary artery disease, angina pectoris, uncontrolled hypertension, serious arrythmias or myocardial infarction within the previous six months.
* Evidence of active infection requiring antibiotic therapy.
* Active intracranial metastases. Patients with previously resected intracranial disease and/or previously irradiated intracranial metastases that have been stable for four weeks are eligible.
* Pregnant or lactating women. Pregnant women are excluded from this study. Women of childbearing potential must have a negative pregnancy test. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated on study.
* Patients requiring systemic corticosteroids (unless patient has had NO STEROIDS IN THE PAST 4 WEEKS).
* Autoimmune disease including, but not limited to, rheumatoid arthritis, systemic lupus erythematous, multiple sclerosis, or ankylosing spondylitis
* Patient must not have post-obstructive pneumonia or other serious infection at the time of registration or other serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
* Subject is not a candidate for complete resection of the carcinoma via pneumonectomy, lobectomy, bilobectomy, extended wedge resection or anatomic segmentectomy with or without sleeve resection as noted in the surgical plan..
* Prior resection of lung cancer is allowed, if at least five years have elapsed between previous resection and registration.
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the patient has been disease-free for at least 5 years prior to registration.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility; patients will be observed for treatment-related toxicity during and after each immunization,and for 1 h after immunization in the event that an immediate-type hypersensitivity reaction occurs. | 2.5 years

SECONDARY OUTCOMES:
To evaluate the ability of the DNA-based vaccine to induce immune responses to the autologous tumor (if available) and/or the vaccine. | 14

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Socinski, MD, Principal Investigator — UPCI/UPMC: Director, Lung Cancer Section, Division of Hematology/Oncology
Locations (2):
- United States (2):
  - University of Pittsburgh Cancer Institute - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania